CLINICAL TRIAL: NCT07329907
Title: Comparative Efficacy of Topical Salicylic Acid/Lactic Acid, Intralesional Candida Antigen, and Their Combination in the Treatment of Warts: A Randomized, Assessor-Blinded, Controlled Trial
Brief Title: Combination Therapy for Warts: Candida Antigen vs. Topical Keratolytic
Acronym: CA-SA/LA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Shams, Principal investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Combination therapy for warts
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Warts; Human Papilloma Virus (HPV)
Keywords: warts; verruca; candida antigen; intralesional immunotherapy; salicylic acid; lactic acid
MeSH Terms: conditions — Warts | interventions — lactic acid, salicylic acid drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor-Blinded (Outcome Assessor Only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- topical monotherapy (Active Comparator): Patients receive topical application of Salicylic Acid 40% and Lactic Acid 16% once daily for up to 6 weeks.
  Interventions: Drug: Salicylic Acid/Lactic Acid Topical Solution
- Intralesional Monotherapy (Active Comparator): Patients receive intralesional injection of Candida Antigen (0.1-0.3 mL) every 2 weeks for up to 6 sessions.
  Interventions: Biological: Candida Antigen Intralesional Injection
- Combination Therapy (Active Comparator): Patients receive intralesional injection of Candida Antigen (0.1-0.3 mL) every 2 weeks for up to 6 sessions, with topical Salicylic Acid 40% and Lactic Acid 16% applied in between.
  Interventions: Combination Product: Candida Antigen and Salicylic Acid/Lactic Acid

INTERVENTIONS:
Drug: Salicylic Acid/Lactic Acid Topical Solution — Patients receive topical application of Salicylic Acid 40% and Lactic Acid 16% once daily for up to 6 weeks.
  Arms: topical monotherapy
Biological: Candida Antigen Intralesional Injection — Patients receive intralesional injection of Candida Antigen (0.1-0.3 mL) every 2 weeks for up to 6 sessions.
  Arms: Intralesional Monotherapy
Combination Product: Candida Antigen and Salicylic Acid/Lactic Acid — Patients receive intralesional injection of Candida Antigen (0.1-0.3 mL) every 2 weeks for up to 6 sessions, with topical Salicylic Acid 40% and Lactic Acid 16% applied in between.
  Arms: Combination Therapy

SUMMARY:
Objective: To compare the efficacy, safety, and recurrence rates of topical salicylic acid/lactic acid (SA/LA) monotherapy (Group A), intralesional Candida antigen (CA) monotherapy (Group B), and their combination (Group C) for the treatment of warts.

ELIGIBILITY:
Inclusion Criteria:

1. Single or multiple warts.
2. Aged 5 to 60 years.
3. Eligible for both topical and intralesional treatments.
4. No prior wart treatment for at least 1 month.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Immunosuppression or use of immunosuppressive drugs.
3. Known sensitivity to study ingredients.
4. Systemic/local inflammation or infection.
5. History of bleeding/clotting disorder, or use of anticoagulants/NSAIDs.
6. History of asthma, allergic skin disorders, or convulsions.
7. History of chronic systemic diseases (renal/hepatic failure, cardiovascular disorders).

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | 3 months post-treatment
  Percentage of patients achieving complete disappearance of all warts.

SECONDARY OUTCOMES:
Distant Wart Clearance Rate | 3 months post-treatment
  Percentage of patients achieving clearance of non-injected/distant warts.
Recurrence Rate | 6 months post-treatment
  Percentage of patients with recurrence of warts after achieving CR.
Safety and Tolerability Profile | At each visit (every 2 weeks) and 3 months post-treatment
  Incidence and severity of local (pain, edema, crustations) and systemic (flu-like symptoms) side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Shams, Principal Investigator — Benha University
Locations (1):
- Outpatient Clinic of Dermatology, Venereology and Andrology Department at Benha University Hospitals, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided